CLINICAL TRIAL: NCT03150498
Title: A Phase 1 Cross-over Study to Determine Food Effects on the Pharmacokinetics of Oral BTD-001 and Metabolites in Healthy Volunteers, Followed by an Optional Multiple Dose Study to Assess Pharmacokinetics of Oral BTD-001
Brief Title: A Food Effects Study and Optional Multi Dose Study to Assess PK of BTD-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Balance Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BTD-001 HV104
Record Dates: First submitted 2017-05-02; First posted 2017-05-12 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Food Effect; Healthy
Keywords: Food Effect; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BTD-001 (fed) (Experimental)
  Interventions: Drug: BTD-001
- BTD-001 (fasted) (Experimental)
  Interventions: Drug: BTD-001

INTERVENTIONS:
Drug: BTD-001 — BTD-001 in fed vs fasted state

SUMMARY:
This is a single-centre, open-label study in healthy male and non-pregnant, non-lactating females. The study will consist of up to 2 parts; the decision to proceed to the optional second part will be made following review of Part 1 data.

Part 1 is a single dose, two period crossover to assess food affect of oral BTD-001.

Optional Part 2 is a non-randomised, single arm study multi dose design to evaluate PK profile of BTD-001

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and non-pregnant, non-lactating females aged 18-55 years old
* BMI between18.0-35.0 kg/m2 unless investigator deems not clinically significant
* Provide written consent
* Agrees to protocol specified contraception

Exclusion Criteria:

* Received any investigational treatment within last 3 months
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week
* Current smokers and those who have smoked, including nicotine replacement or e-cigarates within the last 12 months.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
* Clinically significant abnormal lab results
* Positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Evidence of renal impairment at screening
* History of or current seizure disorder or history of syncope, unexplained loss of consciousness or seizure in the past 3 years
* Clinically significant medical/psychiatric history findings, or physical/neurological examination findings or significant history of or current suicidal ideation or behaviour
* History of or current significant pulmonary, cardiac, renal, hepatic, chronic respiratory, gastrointestinal, neurological or psychiatric disease, substance dependence, porphyria, malignancy (with exception of local cutaneous squamous or basal cell carcinomas or local cervical squamous cell cancer resolved after resection) or hypothyroidism
* Subjects with QT interval corrected for heart rate according to Fridericia's formula of >430 msec in males and >450 msec in females
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
* Donation or loss of greater than 400 mL of blood within the previous 3 months Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than up to 4 g per day paracetamol,hormone replacement therapy and hormonal contraception) or herbal remedies
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Part 1 & Part 2 - Cmax of BTD-001 and major metabolites | [Maximum 30 days]
  Maximum Observed Plasma Concentration
Part 1 & Part 2 - Tmax of BTD-001 and major metabolites | [Maximum 30 days]
  Time to Maximum Observed Plasma Concentration
Part 1 & Part 2 - AUC(0-last): of BTD-001 and major metabolites | [Maximum 30 days]
  Area Under the Curve for Observed Plasma Concentration
Part 1 & Part 2 - T1/2 of BTD-001 and major metabolites | [Maximum 30 days]
  elimination half-life

SECONDARY OUTCOMES:
Physical Examination | [Maximum 30 days]
  Safety and tolerability of BTD-001 by assessing physical examination
Vital Signs | [Maximum 30 days]
  Safety and tolerability of BTD-001 by assessing vital signs
ECG | [Maximum 30 days]
  Safety and tolerability of BTD-001 by assessing ECG
Adverse Events | [Maximum 30 days]
  Safety and tolerability of BTD-001 by assessing AEs
Safety Lab Test | [Maximum 30 days]
  Safety and tolerability of BTD-001 by assessing safety lab tests
Likert Scales | [Maximum 30 days]
  To assess BTD-001 withdrawal in healthy volunteers

OTHER OUTCOMES:
Karolinska Sleepiness Scale | [Maximum 30 days]
  To assess sleepiness using the KSS

CONTACTS AND LOCATIONS:
Overall Officials: Nand Signh, MD, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided